CLINICAL TRIAL: NCT01317368
Title: The Analgesic Effect of Transversus Abdominis Plane (TAP) Block Versus Wound Infiltration Versus Placebo Following Open Radical Prostatectomy, a Double Blinded, Randomized Clinical Trial
Brief Title: The Analgesic Effect of Transversus Abdominis Plane (TAP) Block Following Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Birgitte Ruhnau, Consultant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-AS-2010; 2010-024153-36 (EudraCT Number)
Record Dates: First submitted 2011-03-11; First posted 2011-03-17 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Postoperative Pain
Keywords: Postoperative analgesic treatment; TAP block; Prostatectomy; Double blinded randomized clinical trial
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TAP block (Active Comparator): TAP block with Ropivacaine
  Wound infiltration with Saline
  Interventions: Drug: Naropine
- Wound infiltration (Active Comparator): TAP block with Saline.
  Wound infiltration with Ropivacaine.
  Interventions: Drug: Naropine
- Placebo (Placebo Comparator): TAP block with Saline.
  Wound infiltration with Saline.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naropine — 20 mL of 0,75% Naropin is deposited on each side (40 mL in total) in the TAP.
  At the same time 40 mL of saline 0,9% will be deposited subcutaneously as wound infiltration.
  Both procedures is carried out at the end of the surgery while the patient is still anaesthetized and only this once.
  Other Names: Ropivacaine; TAP block; Wound infiltration; Placebo
  Arms: TAP block
Drug: Naropine — 20 mL Saline 0,9% is deposited on each side (40 mL in total) in the TAP.
  At the same time 40 mL Ropivacaine 0,75% will be deposited subcutaneously as wound infiltration.
  Both procedures is carried out at the end of the surgery while the patient is still anaesthetized and only this once.
  Other Names: Ropivacaine; TAP block; Wound infiltration; Placebo
  Arms: Wound infiltration
Other: Placebo — 20 mL 0,9% Saline is deposited on each side (40 mL in total) in the TAP.
  At the same time 40 mL Saline 0,9% will be given as wound infiltration.
  Both procedures is carried out at the end of the surgery while the patient is still anaesthetized and only this once.
  Other Names: Ropivacaine; TAP block; Wound infiltration
  Arms: Placebo

SUMMARY:
This study is conducted to evaluate different analgesic treatments effect following operation where the prostate gland is surgically removed.

The different treatments the investigators wish to investigate is:

1. Transversus Abdominis Plane (TAP) block.

   The TAP block is a rather new method, where a local anaesthetic is deposited between the two inner abdominal muscles. Between these muscles, the nerves that innervates the anterior part of the abdominal wall is situated.
2. Wound infiltration

   In this method you deposit a local anaesthetic in the edges of the wound.
3. Placebo

No active local treatment is given.

All patients who wish to participate will be allocated to one of three different treatment groups.

Group 1:

Will receive TAP block with a local anaesthetic and wound infiltration with saline.

Group 2:

Will receive wound infiltration with a local anaesthetic and TAP block with saline.

Group 3:

Will receive TAP block with saline and wound infiltration with saline.

Beside this local treatment all patients will be given systemic Paracetamol (tablet) and Ibuprofen (tablet).

In addition all patients will be given a pump containing morphine. The pump is connected to a button which the patient can activate when they experience pain. This enables the patient to control how much morphine he needs, following the operation.

The hypothesis is that the TAP block is superior in reducing pain and thereby reducing morphine consumption compared to wound infiltration and placebo.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 18 and < 35
* Patients who have given their informed consent and have fully understood the nature and limitations of the study
* Patient who is planned for radical prostatectomy

Exclusion Criteria:

* Not able to cooperate to complete the study
* Is not able to speak and understand danish
* Allergy towards the drugs which is used in the study
* Daily use of strong opioids
* Infection at the injection area

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
A mean visual analogue scale (VAS) pain score 4 hours after surgery when moving from a supine to sitting position between the group receiving active TAP block and the placebo group. | 4 hours postoperative

SECONDARY OUTCOMES:
VAS pain score at rest, recorded as a Area Under Curve (AUC/24h) | Recorded 0-24 hours postoperative
  This outcome is assessed 1, 2, 4, 6, 8, 20 and 24 hours postoperative, while the patient is supine in his bed.
  This outcome is recorded in and compared between all three groups.
VAS pain score when moving from a supine to a sitting position, recorded as a Area under Curve (AUC/24h) | Recorded 0-24 hours postoperative
  This outcome is assessed 1, 2, 4, 6, 8, 20 and 24 hours postoperative. This outcome is recorded in and compared between all three groups.
Nausea | Recorded 0-24 hours postoperative
  On a scale ranging none-mild-moderate-severe at 1, 2, 4, 6, 8, 20, 24 hours postoperative.
  This outcome is recorded in and compared between all three groups
Sedation | Recorded at 0-24 hours postoperative
  On a scale ranging none-mild-moderate-severe this outcome is assessed at 1, 2, 4, 6, 8, 20 and 24 hours postoperative.
  This outcome is recorded in and compared between all three groups.
Vomiting | Recorded 0-24 hours postoperative
  The number of times the patient produces more than 10 mL of vomit. Recorded at the intervals 0-1, 1-2, 2-4, 4-6, 6-8, 8-20 and 20-24 hours postoperative This outcome is recorded in and compared between all three groups
On-going morphine consumption | Recorded 0-24 postoperative
  Recorded at the intervals 0-1, 1-2, 2-4, 4-6, 6-8, 8-20 and 20-24 hours postoperative This outcome is recorded and compared between all three groups
Cumulated morphine consumption | 24 hours postoperative
  This outcome is recorded in and compared between all three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Ruhnau, Consultant, Principal Investigator — Department of Anaesthesiology, Abdominal Centre, Rigshospitalet
Locations (1):
- The Department of Anaesthesiology, Abdominal Centre, Rigshospitalet, Copenhagen Ø, Denmark